CLINICAL TRIAL: NCT04469504
Title: Prehabilitaion Program for Sarcopenic Patients Prior to Pancreaticoduodenectomy for Periampullary Malignant Tumors
Brief Title: Preoperative Prehabilitation for Sarcopenic Patients Prior to Pancreatic Surgery for Cancer
Acronym: PSOAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other); Santelys Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2017_06; 2019-A00632-55 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenia; Pancreatic Cancer
Keywords: morbimortality; Prehabilitaion; pancreatic surgery; cephalic duodenopancreatectomy
MeSH Terms: conditions — Sarcopenia; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREHAB (Experimental)
  Interventions: Other: Prehabilitation program
- control group (Active Comparator)
  Interventions: Dietary Supplement: Oral Impact

INTERVENTIONS:
Other: Prehabilitation program — 4-week trimodal prehabilitation program: Exercise, nutritional supplementation, and psychological support
  Arms: PREHAB
Dietary Supplement: Oral Impact — perioperative immunonutrition by ORAL IMPACT
  Arms: control group

SUMMARY:
Major digestive surgery is associated with a significant rate of postoperative complications. To improve postoperative outcome, efforts are focused on postoperative course leading to the concept of rehabilitation. However, the rehabilitation concept does not allow to improve muscular and functional reserves at the time of surgery. Sarcopenia is a condition characterized by loss of skeletal muscle mass and function. Also, the prevalence of sarcopenia in patients with cancer is high and has a prevalence of around 25% in patients with pancreatic cancer, with a considerable impact on postoperative and survival outcomes.

The hypothesis is the preoperative management of sarcopenia by a rehabilitation program could improve patients' operative outcomes by reducing the rate of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy for cancer
* Sarcopenic status

Exclusion Criteria:

* Age younger than 18 years
* Medical contraindications including cardiovascular disease or clinically significant vascular disease
* Physical inability to exercise
* Emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative severe pancreatic fistula (Grade B and C) | at 90 days
  Pancreatic fistula as defined by the International Study Group of pancreatic Fistula (ISGPF)

SECONDARY OUTCOMES:
Rate of Severe postoperative complications | at 90 days
  Grade > IIIa (Clavien-Dindo classification)
Overall survival | at 1 year and at 3 years
Program acceptance measure by Modified ACCEPT© questionnaire | at 30 days
Rate of program completion | at 30 days
  self questionnaire to measure opinion with respect of rehabilitation program
Satisfaction questionnaire by EVAN-G | at 30 days
  EVAN-G general patient satisfaction questionnaire consisting of 26 items divided into 6 sub-sections scoring on a scale from 0 to 100. It is designed to report perioperative problems.
Satisfaction questionnaire by the questionnaire for satisfaction of hospitalized (QSH-45) | at 30 days
  French self-administered instrument for measuring hospitalized patients' satisfaction based on the patient's point of view. QSH contained 45 items describing 9 dimensions, leading to 2 composite scores (staff and structure index)
Quality of life by EORTC-QLQc30 scale | at 1 month, 3 months, 6 months and at 1 year
  The QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The questionnaire includes one global health status/QoL scale, five functional scales and three symptom scale. Each scale is scored from 0 to 100. A high score on a scale indicate a good outcome for the dimension of QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi ELAMRANI, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France